CLINICAL TRIAL: NCT05157204
Title: Measurment of Interleuukin-6 at Exhaled Breath of Condensate of Covid-19 Patients and Post Covid-19 Patients With Lung Fibrosis Randomized Controlled Study
Brief Title: Measurment of Interleuukin-6 at Exhaled Breath Condensate of Covid-19 Patients and Post Covid-19 Patients With Lung Fibrosis Randomized Controlled Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ministry of Health, Saudi Arabia (Other Government)
Responsible Party: Principal Investigator, Amr kamel khalil Ahmed, Saudia Arabia , Riyadh . public health , First health cluster, Ministry of Health, Saudi Arabia
Other Study IDs: saudia arabia
Record Dates: First submitted 2021-12-11; First posted 2021-12-14 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Inflammatory Response; Immunological Abnormality; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- adult 20 patients with moderate to severe covid-19: adult 20 covid-19 patients with moderate to severe covid-19. for measurment of interleukin-6 from exhaled condensate during first 10 days of postive PCR
  Interventions: Procedure: measurment of interleukin-6 at exhaled condensate
- 20 healthy controls adult non pregnant humans f: 20 healthy adults above 18 years non pregnant for measurment of interleukin-6 from exhaled condensate
  Interventions: Procedure: measurment of interleukin-6 at exhaled condensate
- adult 20 patients with moderate to severe postcovid-19: adult 20 post covid-19 patients with moderate to severe covid-19 for measurment of interleukin-6 from exhaled condensate
  Interventions: Procedure: measurment of interleukin-6 at exhaled condensate

INTERVENTIONS:
Procedure: measurment of interleukin-6 at exhaled condensate — the breath condensate samples were collected using a specially designed condensing chamber ( Ecoscreen; Jaeger, Hoechberg, Germany) to measure the interleukin-6 at exhaled condensate of 60 participants

SUMMARY:
COVID-19 has emerged as a global pandemic. It is mainly manifested as pneumonia which may deteriorate into severe respiratory failure. The major hallmark of the disease is the systemic inflammatory immune response characterized by Cytokine Storm (CS). CS is marked by elevated levels of inflammatory cytokines, mainly interleukin-6 (IL-6), IL-8, IL-10, tumour necrosis factor-α (TNF-α) and interferon-γ (IFN-γ). Of these, IL-6 is found to be significantly associated with higher mortality. IL-6 is also a robust marker for predicting disease prognosis and deterioration of clinical profile. (1) IL-6 was detectable in the breath condensate of all the healthy non-smokers, but was significantly higher in the COPD patient. Exhaled breath condensate is totally non-invasive and highly acceptable to patients. The collection procedure has no effect on airway function or inflammation, and there is growing evidence that abnormalities in condensate composition may reflect biochemical changes in airway lining fluid. This method has been successfully used in previous studies to investigate several inflammatory markers in COPD and asthmatic patients. (2) Il-6 is produced in the lung by interstitial fibroblasts, alveolar macrophages, and large-vessel and bronchial epithelial cells. IL-6 levels are high in chronic inflammatory conditions of the lung, such as those due to allogeneic transplantation, bleomycin-induced fibrosis and a variety of human interstitial lung diseases. High levels of IL-6 have been found in the induced sputum of patients with COPD, particularly during exacerbation. Park et al. found increased IL-6 levels in the Bronchioalveolar lavage fluid of patients with non-specific interstitial pneumonia/fibrosis and in some patients with interstitial pneumonia. (3) the study involved 20 healthy controls and 20 patients with moderate to severe covid-19 according to cdc classifaction and 20 patients post covid-19 with lung fibrosis to estimate the measurment of interleukin-6 at exhaled condensate, this clinical randomized control study consists of 3 arms for 6 month ( all participants above 18 years non prgnant humans )

DETAILED DESCRIPTION:
COVID-19 has emerged as a global pandemic. It is mainly manifested as pneumonia which may deteriorate into severe respiratory failure. The major hallmark of the disease is the systemic inflammatory immune response characterized by Cytokine Storm (CS). CS is marked by elevated levels of inflammatory cytokines, mainly interleukin-6 (IL-6), IL-8, IL-10, tumour necrosis factor-α (TNF-α) and interferon-γ (IFN-γ). Of these, IL-6 is found to be significantly associated with higher mortality. IL-6 is also a robust marker for predicting disease prognosis and deterioration of clinical profile. (1) IL-6 was detectable in the breath condensate of all the healthy non-smokers, but was significantly higher in the COPD patient. Exhaled breath condensate is totally non-invasive and highly acceptable to patients. The collection procedure has no effect on airway function or inflammation, and there is growing evidence that abnormalities in condensate composition may reflect biochemical changes in airway lining fluid. This method has been successfully used in previous studies to investigate several inflammatory markers in COPD and asthmatic patients. (2) Il-6 is produced in the lung by interstitial fibroblasts, alveolar macrophages, and large-vessel and bronchial epithelial cells. IL-6 levels are high in chronic inflammatory conditions of the lung, such as those due to allogeneic transplantation, bleomycin-induced fibrosis and a variety of human interstitial lung diseases. High levels of IL-6 have been found in the induced sputum of patients with COPD, particularly during exacerbation. Park et al. found increased IL-6 levels in the Bronchioalveolar lavage fluid of patients with non-specific interstitial pneumonia/fibrosis and in some patients with interstitial pneumonia. (3) Dowlati et al. have reported increased levels of IL-6 in the serum and BAL fluid of patients with lung cancer. (4) A recent study by Bhowmik et al. found increased IL-6 and IL-8 levels in the sputum of COPD patients with frequent exacerbations. (5) Also, at another study Exhaled interleukin-6 and leukotriene B4 levels may be useful noninvasive markers of airway inflammation in cigarette smokers. (6) These studies and our novel method after clinical trials may open the field for future therapies for covid-19 and post covid-19 lung fibrosis by inhaler transport medicines as a new challenge for overcome sequels of this pandemic. And this suggested new procedure for measurement of exhaled il-6 take us to study which is IL-6 is risky is IL-6 produced from airway or endocrine IL-6 or immune IL-6 From previous studies we need a procedure acceptable to patients and easy, noninvasive, sensitive he study involved 20 healthy controls and 20 patients with moderate to severe covid-19 according to cdc classifaction and 20 patients post covid-19 with lung fibrosis to estimate the measurment of interleukin-6 at exhaled condensate, this clinical randomized control study consists of 3 arms for 6 month ( all participants above 18 years non prgnant humans )

ELIGIBILITY:
Inclusion Criteria:

* age above 18 years
* covid-19 patients (20) with real time PCR positive test moderate to severe according to CDC classification
* smokers are included
* post-covid 19 patients with real-time pcr positive test
* 20 healthy subjects

Exclusion Criteria:

* below 18 years and above 80 years pregnant womens any medications as anti-il-6 unstable cases history of copd cases or lung disease or lung cancer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: the partcipants are 60 human subjects divided to 3 arms 20 healthy subjects 20 covid-19 patients with new real time PCR positive and during first 10 days of result 20 postcovid-19 patients with lung fibrosis and also current real time PCR positive all subjects have informed consent
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-01-26 (Estimated); Primary Completion 2022-04-26 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
measurement of interleukin-6 at exhaled condensate in covid-19, postcovid-19 ,healthy subjects | 6 month

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol